CLINICAL TRIAL: NCT01876472
Title: Differences in Music Perception Skills Between Child, Teen and Adult Cochlear Implant Recipients
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: VD_2011_11_15
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-05

CONDITIONS: Cochlear Implant Recipients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Children aged 3 - 10 years: Assessment of music perception skills with cochlear implant recipients aged 3 - 10 years
  Interventions: Behavioral: Assessment of music perception skills
- Teenagers aged 11 - 15 years: Assessment of music perception skills with cochlear implant recipients aged 11 - 15 years
  Interventions: Behavioral: Assessment of music perception skills
- Adults aged 16 - 70 years: Assessment of music perception skills with cochlear implant recipients aged 16 - 70 years
  Interventions: Behavioral: Assessment of music perception skills

INTERVENTIONS:
Behavioral: Assessment of music perception skills — A sequence of tones is presented to participants. Then the same sequence is presented again, with the 4th tone being one to six half tones different from the first sequence. Participants are asked to indicate when they hear a difference betweent the first and the second sequence.

SUMMARY:
Adult recipients of cochlear implants (CI) generally loose interest in listening to music. This may be due to the rather limited spectral resolution of CI. However, child CI-recipients, if offered the opportunity, like to listen to music. They participate actively in musical acitivities, such as singing, dancing or playing an instrument. Thus, there seems to be a fundamental difference in the music perception of people who receive CI as child or as adult.

This study assesses music perception skills of child, teen and adult cochlear implant recipients in settings with simple tone sequences and in a more complex, melodious context.

ELIGIBILITY:
Inclusion criteria:

* Participants are uni- or bilateral CI recipients.
* Participants are at least 3 years old.
* Participants received CI one or more years before.
* Participants are healthy.
* Participation in the study is voluntary.
* Participants and their legal custodians have read the information for participants at least one day prior to the test and given their written consent.

Exclusion criteria:

* Surgery for CI carried out less than one year before the test.
* Children less than 3 years old.
* Reduced cognitive capabilities due to old age.
* Physical or mental handicaps.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Healthy CI recipients that receive their regular follow-ups in the ENT-clinic of the Zurich University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Does the age at which a person receives a cochlear implant influence music perception skills? | Test and retest are taken within 6 months
  The test assesses wether cochlear implant carriers are able to hear the difference betweent two sequences of sounds, where in the second sequence on tone is different from the first sequence. If a difference is perceived, then the test assesses how big this difference has to be in order to be heard.
  The first and the second test are no more than six months apart; both times the same procedure is followed.
  The test is carried out with three age groups:
  1. Children aged 3-10 years
  2. Teenagers aged 11 - 14 years
  3. Persons above 15 years

SECONDARY OUTCOMES:
Do the results of the primary outcome measure depend on the tone sequence presented to the cochlear implant recipients? | Test and retest are no more than 6 months apart
  The test is carried out with three different tone sequences:
  1. Same tone at three different octaves (control tune: 131 Hz, 262 Hz, 523 Hz)
  2. Tune of rising, then falling notes
  3. Tune of rising notes only

OTHER OUTCOMES:
How can the findings of the primary and the secondary outcome measure be used to improve music perception with existing cochlear implants? | 6 months
  Can the results of the primary and the secondary outcome measure be applied to improve music perception with existing cochlear implants - e.g. by changing / adapting algorithms?

CONTACTS AND LOCATIONS:
Overall Officials: Dorothe Veraguth, MD, Principal Investigator — University Hospital Zurich, Clinic for Otorhinolaryngology
Locations (1):
- University Hospital Zurich,, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Svirsky MA, Robbins AM, Kirk KI, Pisoni DB, Miyamoto RT. Language development in profoundly deaf children with cochlear implants. Psychol Sci. 2000 Mar;11(2):153-8. doi: 10.1111/1467-9280.00231. PMID 11273423
- [Background] Nicholas JG, Geers AE. Effects of early auditory experience on the spoken language of deaf children at 3 years of age. Ear Hear. 2006 Jun;27(3):286-98. doi: 10.1097/01.aud.0000215973.76912.c6. PMID 16672797
- [Background] Svirsky MA, Teoh SW, Neuburger H. Development of language and speech perception in congenitally, profoundly deaf children as a function of age at cochlear implantation. Audiol Neurootol. 2004 Jul-Aug;9(4):224-33. doi: 10.1159/000078392. PMID 15205550
- [Background] Fujita S, Ito J. Ability of nucleus cochlear implantees to recognize music. Ann Otol Rhinol Laryngol. 1999 Jul;108(7 Pt 1):634-40. doi: 10.1177/000348949910800702. PMID 10435919
- [Background] Green T, Faulkner A, Rosen S. Spectral and temporal cues to pitch in noise-excited vocoder simulations of continuous-interleaved-sampling cochlear implants. J Acoust Soc Am. 2002 Nov;112(5 Pt 1):2155-64. doi: 10.1121/1.1506688. PMID 12430827
- [Background] Peretz I, Hyde KL. What is specific to music processing? Insights from congenital amusia. Trends Cogn Sci. 2003 Aug;7(8):362-367. doi: 10.1016/s1364-6613(03)00150-5. PMID 12907232
- [Background] Fitzsimons M, Sheahan N, Staunton H. Gender and the integration of acoustic dimensions of prosody: implications for clinical studies. Brain Lang. 2001 Jul;78(1):94-108. doi: 10.1006/brln.2000.2448. PMID 11412018
- [Background] Shannon RV, Zeng FG, Kamath V, Wygonski J, Ekelid M. Speech recognition with primarily temporal cues. Science. 1995 Oct 13;270(5234):303-4. doi: 10.1126/science.270.5234.303. PMID 7569981
- [Background] K. Gfeller, S. A. Witt, L. J. Spencer, J. Stordahl and B. Tomblin (1999), Musical Involvement and Enjoyment of Children Who Use Cochlear Implants, Volta Review, 100(4), pp. 213-233
- [Background] Mitani C, Nakata T, Trehub SE, Kanda Y, Kumagami H, Takasaki K, Miyamoto I, Takahashi H. Music recognition, music listening, and word recognition by deaf children with cochlear implants. Ear Hear. 2007 Apr;28(2 Suppl):29S-33S. doi: 10.1097/AUD.0b013e318031547a. PMID 17496641
- [Background] Cooper WB, Tobey E, Loizou PC. Music perception by cochlear implant and normal hearing listeners as measured by the Montreal Battery for Evaluation of Amusia. Ear Hear. 2008 Aug;29(4):618-26. doi: 10.1097/AUD.0b013e318174e787. PMID 18469714
- [Background] Sharma A, Dorman MF, Kral A. The influence of a sensitive period on central auditory development in children with unilateral and bilateral cochlear implants. Hear Res. 2005 May;203(1-2):134-43. doi: 10.1016/j.heares.2004.12.010. PMID 15855038
- [Background] Looi V, She J. Music perception of cochlear implant users: a questionnaire, and its implications for a music training program. Int J Audiol. 2010 Feb;49(2):116-28. doi: 10.3109/14992020903405987. PMID 20151886
- [Background] Gfeller K, Turner C, Mehr M, Woodworth G, Fearn R, Knutson JF, Witt S, Stordahl J. Recognition of familiar melodies by adult cochlear implant recipients and normal-hearing adults. Cochlear Implants Int. 2002 Mar;3(1):29-53. doi: 10.1179/cim.2002.3.1.29. PMID 18792110
- [Background] Trehub SE, Cohen AJ, Thorpe LA, Morrongiello BA. Development of the perception of musical relations: semitone and diatonic structure. J Exp Psychol Hum Percept Perform. 1986 Aug;12(3):295-301. doi: 10.1037//0096-1523.12.3.295. PMID 2943857